CLINICAL TRIAL: NCT00729924
Title: Genetic Predictors of Raltegravir Penetration Into Cerebrospinal Fluid
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, David Haas, Professor of Medicine, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 080536
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Results first posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: Raltegravir; CSF; ABCB1 SNP; HIV/AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label oral raltegravir (Experimental): Raltegravir a single 400 mg pill taken orally every 12 hours for a total of 7 days.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — 400mg orally every 12 hours for 7 days
  Other Names: MK-0518

SUMMARY:
This study is being done to find out how much of the drug raltegravir (RGV) gets into cerebrospinal fluid (CSF), compared to how much get into the blood and to find out if normal changes in a certain gene in your body affects how much RGV gets into the CSF.

DETAILED DESCRIPTION:
The multidrug efflux transporter P-glycoprotein (P-gp) is expressed in the blood-brain barrier where it limits entry of substrate drugs into the central nervous system. Raltegravir (MK-0158), a new HIV-1 integrase inhibitor and potentially major addition to the therapeutic armamentarium against HIV, is a substrate for P-gp. Studies are warranted to elucidate the relevance of P-gp transport for raltegravir in the central nervous system.

ELIGIBILITY:
Inclusion criteria:

1. Able to give informed consent.
2. Negative HIV-1 serology.
3. At least 18 but no more than 55 years of age.
4. Body mass index <30.
5. Estimated creatinine clearance ≥ 50 mL/minute within 30 days prior to study entry.
6. Within 30 days prior to study entry:

   * Absolute neutrophil count ≥ 1,000/mm3.
   * Hemoglobin ≥ 12.5 g/dL for males and ≥ 11.5 g/dL for females.
   * Platelet count ≥ 100,000/mm3.
   * AST, ALT, and total bilirubin within normal range.
   * Alkaline phosphatase < or = 1.5 x upper limit of normal.
7. Female study volunteers of reproductive potential must have a negative serum or urine pregnancy test performed within 30 days before study entry.
8. Must agree not to participate in a conception process.
9. Drug transporter gene ABCB1 position 3435 genotype C/C or T/T.

Exclusion criteria:

1. Use of any medication that is metabolized by CYP3A or UGT1A1.
2. Anticipated need to take any medication that is metabolized by CYP3A or UGT1A1 during the study.
3. Active drug use or dependence.
4. Inability to abstain from alcohol-containing beverages, grapefruit, and grapefruit juice.
5. Serious illness that would interfere with study participation.
6. Hospitalization for any reason or therapy for serious illness within 14 days prior to study entry.
7. History of hypersensitivity to study drug or its formulation.
8. As determined by the investigator, a significant active or previous history of cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, or immunologic disease(s). This is inclusive of chronic illnesses such as hypertension, coronary artery disease, arthritis, diabetes, any chronic gastrointestinal conditions that may affect drug absorption, etc.
9. Breast-feeding.
10. Evidence of CNS infection or space occupying lesion by history or physical examination.
11. History of significant CNS disorder.
12. Prisoners or subjects who are compulsorily detained.
13. ABCB1 position 3435 C/T heterozygosity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Haas, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Therapeutics Clinical Research Site, Nashville, Tennessee, United States

REFERENCES:
- [Result] Johnson DH, Sutherland D, Acosta EP, Erdem H, Richardson D, Haas DW. Genetic and non-genetic determinants of raltegravir penetration into cerebrospinal fluid: a single arm pharmacokinetic study. PLoS One. 2013 Dec 11;8(12):e82672. doi: 10.1371/journal.pone.0082672. eCollection 2013. PMID 24349334

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir 400mg Orally Every 12 Hours for 7 Days.: Raltegravir a single 400mg tablet taken orally every 12 hours for a total of 7 days.
Period: Overall Study
Arm/Group | Raltegravir 400mg Orally Every 12 Hours for 7 Days.
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Raltegravir: 400mg Orally Every 12 Hours for 7 Days: Raltegravir a single 400mg tablet taken orally every 12 hours for a total of 7 days.
Arm/Group | Raltegravir: 400mg Orally Every 12 Hours for 7 Days
Number analyzed (Participants) | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.5 [26.8 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40
Cerebrospinal Fluid Protein [Median (Inter-Quartile Range); unit: mg/dL] | 33 [24 to 43]
Weight [Median (Inter-Quartile Range); unit: kilograms] | 74.6 [62.6 to 80.5]
Body Mass Index [Median (Inter-Quartile Range); unit: kilgrams/(meter squared)] | 24.0 [22.2 to 25.6]
ABCB1 Genotype [Number; unit: participants] — ABCB1 (rs1045642) C/C or T/T Genotype
  participants
    C/C Genotype | 20
    T/T Genotype | 20

OUTCOME MEASURES:

1. Primary Outcome: Penetration of Raltegravir (RGV) Into Cerebrospinal Fluid (CSF) Based on Plasma Area-under-the-curve.
Description: The primary outcome for this study was the ratio of the 4-hour CSF concentration value (ng/mL) to the partial plasma area-under-the-curve 0-4h value (h*ng/mL).
Time Frame: Day 7
Measure: Median (Inter-Quartile Range); unit: 1/h
Groups:
- Raltegravir: 400mg Orally Every 12 Hours for 7 Days (ABCB1 C/C: Raltegravir a single 400 mg pill taken orally every 12 hours for a total of 7 days in participants with ABCB1 C/C genotype.
- Raltegravir: 400mg Orally Every 12 Hours for 7 Days (ABCB1 T/T: Raltegravir a single 400 mg pill taken orally every 12 hours for a total of 7 days in participants with ABCB1 T/T genotype.
Arm/Group | Raltegravir: 400mg Orally Every 12 Hours for 7 Days (ABCB1 C/C | Raltegravir: 400mg Orally Every 12 Hours for 7 Days (ABCB1 T/T
Number analyzed (Participants) | 20 | 20
1/h | 0.0066 [0.0050 to 0.0081] | 0.0070 [0.0060 to 0.0095]
Statistical Analysis 1: Comparison: Raltegravir: 400mg Orally Every 12 Hours for 7 Days (ABCB1 C/C vs Raltegravir: 400mg Orally Every 12 Hours for 7 Days (ABCB1 T/T; The hypothesis was that the ratio of the 4-hour CSF concentration value to the partial plasma area-under-the-curve 0-4h value would differ between participants with ABCB1 C/C and T/T genotypes; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney) — The p-value is not adjusted for multiple comparisons

2. Secondary Outcome: Penetration of Raltegravir (RGV) Into Cerebrospinal Fluid (CSF) Based on Single Plasma Timepoint.
Description: This outcome was the ratio of the 4-hour CSF concentration value (ng/mL) to the 4-hour plasma concentration value (ng/mL).
Time Frame: Day 7
Measure: Median (Inter-Quartile Range); unit: ratio
Groups:
- Raltegravir: 400mg Orally Every 12 Hours for 7 Days: ABCB1 C/C: Raltegravir a single 400 mg pill taken orally every 12 hours for a total of 7 days in participants with ABCB1 C/C genotype.
- Raltegravir: 400mg Orally Every 12 Hours for 7 Days: ABCB1 T/T: Raltegravir a single 400 mg pill taken orally every 12 hours for a total of 7 days in participants with ABCB1 T/T genotype.
Arm/Group | Raltegravir: 400mg Orally Every 12 Hours for 7 Days: ABCB1 C/C | Raltegravir: 400mg Orally Every 12 Hours for 7 Days: ABCB1 T/T
Number analyzed (Participants) | 20 | 20
ratio | 0.028 [0.014 to 0.057] | 0.021 [0.016 to 0.045]
Statistical Analysis 1: Comparison: Raltegravir: 400mg Orally Every 12 Hours for 7 Days: ABCB1 C/C vs Raltegravir: 400mg Orally Every 12 Hours for 7 Days: ABCB1 T/T; We explored post-hoc whether the ratio of the 4-hour CSF concentration value to the 2-hour plasma concentration differs between participants with ABCB1 C/C and T/T genotypes; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney) — The p-value is not adjusted for multiple comparisons

ADVERSE EVENTS:
Groups:
- Raltegravir: 400mg Orally Every 12 Hours for 7 Days: Raltegravir a single 400 mg pill taken orally every 12 hours for a total of 7 days.
Arm/Group | Raltegravir: 400mg Orally Every 12 Hours for 7 Days
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir: 400mg Orally Every 12 Hours for 7 Days (N=40)
post-lumbar puncture headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitations to this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No